CLINICAL TRIAL: NCT05804851
Title: Skin Microbiome of Chinese Population Cohort Study: Association Between Human Health and Skin Microbiome
Brief Title: Skin Microbiome of Chinese Population Cohort Study
Status: Active, not recruiting | Type: Observational
Sponsor: Westlake University (Other)
Responsible Party: Sponsor
Other Study IDs: 20230103TL001
Record Dates: First submitted 2023-03-23; First posted 2023-04-07 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Skin Microbiome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational study aims to investigate the relationship between public health and the skin microbiome in the province of Zhejiang. Due to the lack of current research on the skin microbiome, the following general questions will be investigated in this study: 1) What connection exists between dietary practices and facial skin microbiome? 2) How do people's lifestyle routines affect the facial skin microbiome? 3) What effects does the altered living environment have on people's facial skin microbiomes? 4) How do the seasons affect people's facial skin microbiomes?

Every 3 to 4 months, the participants' facial skin microbiota samples will be taken, and they will be asked to complete a survey.

ELIGIBILITY:
Inclusion Criteria:

* ages from 10+.

Exclusion Criteria:

* a severe medical history, including a history of surgery or medication, or serious illnesses such as cancer, liver disease, kidney disease, or craniocerebral trauma.
* recent medical treatment (topical antibiotics, corticosteroids, and other anti-inflammatory drugs within 4 weeks, and systemic antibiotics, corticosteroids, and other immunosuppressive drugs within 6 months)

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population of this study will be selected from people that reside in Zhejiang province, and they should fulfill the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in facial microbiota profiling | Day 1, Day 90, Day 180, Day 270, and Day 360
  Quantitative and qualitative analysis of bacteria population from the sample, rRNA and metagenome sequencing will be conducted on each sample

CONTACTS AND LOCATIONS:
Locations (1):
- Westlake University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No